CLINICAL TRIAL: NCT03028311
Title: Feasibility of Single Session In-Room Yttrium-90 Radioembolization Diagnostic Angiography and Treatment
Brief Title: Yttrium Y-90 Radioembolization in Treating Patients With Metastatic Liver Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 2016-0244; NCI-2017-00629 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0244 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Liver Carcinoma; Stage IV Liver Cancer; Stage IVA Liver Cancer; Stage IVB Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Cerebral Angiography; X-Rays; Photons; Technetium Tc 99m Aggregated Albumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (angiography, yttrium Y-90 radioembolization) (Other): The first 2 patients enrolled receive standard of care diagnostic and treatment during 2 visits for approximately 6 hours each within 2-4 weeks. During the first visit, patients undergo diagnostic angiography with embolization of potential hepatoenteric collaterals, receive technetium Tc-99m albumin aggregated as a surrogate to the therapy microspheres via catheter, and undergo planar imaging. During the second visit, patients undergo a second angiography and receive yttrium Y 90 resin microspheres via arterial microcatheter. Patients then undergo single-photon emission computed tomography-computed tomography (SPECT-CT) Bremsstrahlung imaging.
  All subsequent patients enrolled undergo the same previously described diagnostic and treatment during 1 visit over about 8 hours.
  Interventions: Procedure: Angiography; Procedure: Computed Tomography; Procedure: Planar Imaging; Radiation: Radioembolization; Procedure: Single Photon Emission Computed Tomography; Radiation: Technetium Tc-99m Albumin Aggregated; Other: Yttrium Y 90 Resin Microspheres

INTERVENTIONS:
Procedure: Angiography — Undergo angiography
Procedure: Computed Tomography — Undergo SPECT-CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Procedure: Planar Imaging — Undergo planar imaging
Radiation: Radioembolization — Undergo radioembolization
  Other Names: intra-arterial brachytherapy
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT-CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Radiation: Technetium Tc-99m Albumin Aggregated — Given via arterial catheter
  Other Names: Tc 99m-labeled MAA; Technetium Tc 99m-Labeled Macroaggregated Albumin; Technetium Tc-99m Albumin Colloid
Other: Yttrium Y 90 Resin Microspheres — Given via arterial catheter
  Other Names: SIR-Spheres

SUMMARY:
This clinical trial studies the side effects and best way to perform yttrium Y-90 radioembolization in treating patients with liver cancer that has spread to other places in the body (metastatic). Yttrium Y-90 radioembolization is a therapy that injects radioactive microspheres directly into an artery that feeds liver tumors to cut off their blood supply. Performing yttrium Y-90 radioembolization in a single session may make treatment faster, minimize patient travel, and decrease the overall cost of the procedure.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility and safety of same day yttrium-90 radioembolization planning and treatment angiography.

SECONDARY OBJECTIVES:

I. To determine the patient costs associated with same diagnostic and treatment compared when compared to the standard two session methodology.

II. To determine the time required to perform the mandatory in-room technetium Tc-99m albumin aggregated (99mTc-MAA) imaging and the associated calculations for the lung shunt fraction and treatment 90Y-microsphere activity.

III. To determine the time for delivery of the therapy 90Y-microsphere radioactivity to the angiography suite after the therapy written directive by the authorized user.

OUTLINE:

The first 2 patients enrolled receive standard of care diagnostic and treatment during 2 visits for approximately 6 hours each within 2-4 weeks. During the first visit, patients undergo diagnostic angiography with embolization of potential hepatoenteric collaterals, receive technetium Tc-99m albumin aggregated as a surrogate to the therapy microspheres via catheter, and undergo planar imaging. During the second visit, patients undergo a second angiography and receive yttrium Y 90 resin microspheres via arterial microcatheter. Patients then undergo single-photon emission computed tomography-computed tomography (SPECT-CT) Bremsstrahlung imaging.

All subsequent patients enrolled undergo the same previously described diagnostic and treatment during 1 visit over about 8 hours.

After completion of study treatment, patients are followed up at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* The ability to understand and sign informed consent
* Any candidate eligible for standard of care Y90 radioembolization for treatment of their primary or metastatic liver tumors

Exclusion Criteria:

* Patients with greater than 50% liver tumor burden

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Success of same day yttrium Y-90 radioembolization planning and treatment angiography | Up to 6 months
  Success will be defined as treatment dose calculated and patient treated on the same day of initial radiation. Feasibility will be defined as at least 9 successful same day treatments. A procedure lasting greater than 4 hours will be considered a failure. The time associated with various aspects of the same-day yttrium Y-90 radioembolization procedure will be determined. Will determine the time and cost for the patient and for MD Anderson Cancer Center between the same day yttrium Y-90-radioembolization treatment and the current standard of care two-day treatment schedule. Success status will be summarized using frequencies and percentages. Success rate will be estimated along with exact 95% confidence interval. Patient characteristics will be summarized using appropriate summary statistics.
Incidence of adverse event assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 6 months
  The summaries will be overall (severity grades 1 through 5). Actions taken for grade 3 events will also be reported. The summaries will present the number and percentage of patients reporting and adverse event for each classification level as well as the number events reported. Laboratory values will be summarized by the treatment group over time.

CONTACTS AND LOCATIONS:
Overall Officials: Armeen Mahvash, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org